CLINICAL TRIAL: NCT00898768
Title: Capsule Endoscopy in Lynch Syndrome for Small Intestinal Tumor Screening
Brief Title: Capsule Endoscopy to Screen for Small Bowel Neoplasia in Lynch Syndrome
Acronym: CELSIUS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); St. Antonius Hospital (Other); The Netherlands Cancer Institute (Other); University Medical Center Nijmegen (Other); Maastricht University Medical Center (Other); Free University Medical Center (Other); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Jan J Koornstra, dr, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CELSIUS; Dutch Cancer Society 2008-4187
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Lynch Syndrome; Small Bowel Neoplasia
Keywords: Lynch syndrome; HNPCC; Capsule endoscopy; Small bowel cancer; Double balloon endoscopy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy (Other): capsule endoscopie at baseline and after 2 years
  Interventions: Procedure: Capsule endoscopy

INTERVENTIONS:
Procedure: Capsule endoscopy — Capsule endoscopy at baseline and after 2 years
  Other Names: Capsule endoscopy PillCamSB

SUMMARY:
Lynch syndrome (LS), or hereditary nonpolyposis colorectal cancer (HNPCC), is a hereditary disorder characterized by a very high risk of early-onset colorectal and endometrial cancer and an increased risk of other cancers, including cancers of the stomach, ovary, urinary tract, hepatobiliary tract, pancreas and small bowel. This is a national multi-centre study evaluating the yield of small bowel screening using capsule endoscopy (CE) and double balloon enteroscopy (DBE) in Lynch syndrome subjects. The intervention consists of performing a capsule endoscopy procedure at baseline and at 2-year follow-up. In patients with polyps or malignant appearing abnormalities on capsule endoscopy, double balloon enteroscopy will be performed with subsequent endoscopic or surgical removal of neoplastic lesions. The aim of the study is to determine the prevalence and incidence of small bowel neoplasia in Lynch syndrome patients using small bowel CE and DBE.

DETAILED DESCRIPTION:
Lynch syndrome (LS), or hereditary nonpolyposis colorectal cancer (HNPCC), is an autosomal dominantly inherited disorder characterized by a very high risk of early-onset colorectal and endometrial cancer and an increased risk of other cancers, including cancers of the stomach, ovary, urinary tract, hepatobiliary tract, pancreas and small bowel. LS is caused by germline mutations in one of the mismatch repair (MMR) genes, mostly hMLH1, hMSH2 and hMSH6. Recently, several studies, including one from the Netherlands, have evaluated the life-time risk of small bowel cancer (SBC) in LS patients. From these studies the life-time risk of SBC is estimated around 4%. This is similar to the life-time risk of colorectal cancer in the general population, for which screening is generally advised. The risk of SBC increases with age, with an estimated prevalence of 1:500 at the age of 40, rising to an estimated prevalence of around 1:70 at the age of 60. Compared with the general population, LS patients with SBC generally present 10-20 years earlier as most patients with sporadic SBC are in their sixth or seventh decade of life. The localisation of SBC in LS is almost equal in the duodenum and jejunum, with localisation in the ileum generally occurring at a lower frequency.Until now, screening for small bowel neoplasia in Lynch syndrome patients is generally not recommended. However, the development of two new techniques to visualize the small intestine has raised the question whether screening might be useful and advisable. Small bowel capsule endoscopy (CE) has been developed as a safe, patient-friendly, minimally invasive modality for visualization of the small bowel. In addition, double-balloon enteroscopy (DBE) has been developed, a technique which allows endotherapeutic interventions. The diagnostic yields of both techniques are markedly higher than the conventional methods, such as push-enteroscopy and enteroclysis. To date, no study has been performed on screening for small bowel neoplasia in Lynch syndrome patients by means of these techniques.

The primary aim of the study is to determine the prevalence and incidence of small bowel neoplasia in Lynch syndrome patients using small bowel CE and DBE.

Secondary objectives:

The secondary aim is to identify risk factors for small bowel pathology useful in clinical practice to identify patients that might benefit from screening and to determine the additional interventional risk associated with the endoscopic procedures.

This is a national multi-centre study evaluating the yield of small bowel screening using capsule endoscopy and double balloon enteroscopy in Lynch syndrome subjects. The intervention consists of performing a capsule endoscopy procedure at baseline and at 2-year follow-up. In patients with polyps or malignant appearing abnormalities on capsule endoscopy, double balloon enteroscopy will be performed with subsequent endoscopic or surgical removal of neoplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic proven mutation carriers, with a known mutation in the hMLH1, hMSH2 or hMSH6 gene.
2. Age between 35 and 70 years.
3. Written informed consent provided.

Exclusion Criteria:

1. Subjects with a strong suspicion on a small bowel stricture.
2. Subjects with previous small bowel surgery.
3. Pregnancy.
4. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The main outcome measure will be the number of neoplastic small bowel lesions, with determination of size, location and histological characteristics at baseline and at follow-up after 2 years. | At baseline and at 2 years

SECONDARY OUTCOMES:
The secondary endpoint will be the number of complications following endoscopic procedures: rates of capsule retention and postpolypectomy bleeding and perforation. | At baseline and at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Koornstra, MD PhD, Principal Investigator — University Medical Center Groningen; Jan H Kleibeuker, MD PhD, Principal Investigator — University Medical Center Groningen; Hans F Vasen, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Haanstra JF, Al-Toma A, Dekker E, Vanhoutvin SA, Nagengast FM, Mathus-Vliegen EM, van Leerdam ME, de Vos tot Nederveen Cappel WH, Sanduleanu S, Veenendaal RA, Cats A, Vasen HF, Kleibeuker JH, Koornstra JJ. Prevalence of small-bowel neoplasia in Lynch syndrome assessed by video capsule endoscopy. Gut. 2015 Oct;64(10):1578-83. doi: 10.1136/gutjnl-2014-307348. Epub 2014 Sep 10. PMID 25209657